CLINICAL TRIAL: NCT05278052
Title: Standard Maintenance Therapy Versus Local Consolidative Radiation Therapy and Standard Maintenance Therapy in 1-5 Sites of Oligometastatic Non-small Cell Lung Cancer (NSCLC): A Phase III Randomized Controlled Trial
Brief Title: Standard Maintenance Therapy (SMT) vs Local Consolidative Radiation Therapy and SMT in OM-NSCLC
Acronym: TARGET-02
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Anil Tibdewal, Principal Investigator, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3445; CTRI/2020/04/024761 (Registry Identifier: Clinical Trial Registry of India)
Record Dates: First submitted 2022-02-22; First posted 2022-03-14 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Oligometastatic Disease; Metastatic Non Small Cell Lung Cancer
Keywords: Local Consolidative Radiation Therapy; Oligometastatic disease; NSCLC; Maintenance therapy; SABR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Phase III, Open-label, Randomized controlled trial,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A: Standard maintenance therapy alone (Active Comparator): Maintenance systemic therapy/ observation
  Interventions: Drug: Standard maintenance therapy as decided by the treating medical oncologist
- ARM B: Local consolidative radiation therapy (LCRT) (Experimental): Radiation therapy to all oligometastatic sites including primary loco-regional disease
  Interventions: Radiation: Local consolidative radiation therapy; Drug: Standard maintenance therapy as decided by the treating medical oncologist

INTERVENTIONS:
Radiation: Local consolidative radiation therapy — Local consolidative radiation therapy (LCRT) to all oligo-metastatic sites in addition to primary disease site
  Other Names: LCRT
  Arms: ARM B: Local consolidative radiation therapy (LCRT)
Drug: Standard maintenance therapy as decided by the treating medical oncologist — Standard maintenance therapy/Observation

SUMMARY:
Standard Maintenance Therapy versus Local Consolidative Radiation Therapy and standard maintenance therapy in 1-5 sites of OligoMetastatic Non-small cell lung cancer (NSCLC): A Phase III Randomized Controlled Trial

DETAILED DESCRIPTION:
Standard of care maintenance therapy alone (standard arm) versus local consolidative radiation therapy and standard of care maintenance therapy (Experimental arm)

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Patients with ECOG performance status of 0-2
3. Patients with pathologically proven diagnosis of NSCLC
4. Patients with 1-5 sites of metastatic disease not including the primary tumor and regional nodes (less than or equal to 3 metastatic lesions in one organ will be eligible and 4 or more metastatic lesions in one organ will be ineligible)
5. Patients who have received standard duration of systemic therapy (4 - 6 cycles) without progression of the disease
6. Patients suitable for definitive therapy to the primary disease
7. All the Oligometastases lesions should be radiologically visible and suitable for ablative doses of radiation in accordance with the dose fractionation regimens specified in the protocol.
8. Patients who have received ablative radiation therapy or surgery or RFA for metastatic sites at presentation or during systemic therapy will be eligible provided the total number of oligometastatic sites at the time of study entry (treated site included) is less than or equal to five.
9. Patients who have received palliative RT for symptomatic bony metastases or RFA will also be eligible provided the treated site is under control on imaging. If not controlled, could be eligible for study if further ablative doses of radiation can be delivered according to the treating physician.
10. Patients who underwent surgical decompression, or stabilization followed by palliative radiation therapy for bony metastases will be eligible in the study provided the treated site is under control on imaging and patient has less than 5 sites of metastases at the time of study entry.
11. Adequate end organ function CBC/differential obtained within 15 days prior to registration on study, with adequate bone marrow function defined as follows:

    * Absolute neutrophil count (ANC) ≥ 500 cells/mm3;
    * Platelets ≥ 50,000 cells/mm3;
    * Hemoglobin ≥ 8.0 g/dl (Use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable);
12. For females of child-bearing potential, negative serum or urine pregnancy test within 14 days prior to study registration;
13. Patients willing for written informed consent and must be willing to comply with the specified follow up schedule

Exclusion Criteria:

1. Patients with progressive disease after initial standard systemic therapy
2. Patients with oncogene driver mutations
3. Patients with more than 5 sites of oligo metastases
4. Patients with metastatic lesion size of more than 5 cm
5. Patients with more than three metastatic lesion in one organ
6. Patients not suitable for definitive radiation therapy to primary disease
7. Patients not suitable for ablative radiation therapy to metastatic sites
8. Patients with malignant peritoneal disease
9. Patients with malignant pleural effusion
10. Leptomeningeal disease
11. Brain metastases in the brain stem
12. Clinical or radiological evidence of spinal cord compression or metastases within 2 mm of spinal cord on MRI
13. Severe, active co-morbidity defined as follows:

    * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
    * Transmural myocardial infarction within the last 6 months;
    * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration;
14. Patients with prior history of radiation therapy to thorax
15. Patients with previous history of malignancy within last 3 years from the date of diagnosis
16. Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2028-04-20 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Upto 2 years
  Overall survival is defined as the duration between the date of randomization to the date of death due to any cause or the date of last follow-up, whichever is earlier.

SECONDARY OUTCOMES:
Progression free survival (PFS ) | Upto 2 years
  Progression free survival is defined as the duration between the date of randomization to the date of first documented progression or death due to any cause or date of last follow-up, whichever is earlier.
Local control rates of treated sites | Upto 2 years
  Local control rate will be defined as the absence of progressive disease at the treated sites
New distant metastases | Upto 2 years
  Time to onset of new distant metastases
Health Related QOL using the EORTC-QLQ-C30 questionnaire | From randomization every 3 months till 2 years
  To evaluate patient reported outcomes between the two arms
Health Related QOL using the EORTC- LC13 questionnaire | From randomization every 3 months till 2 years
  To evaluate patient reported outcomes between the two arms
Response rates | From randomization every 3 months upto 2 years
  To compare response rates between the two arms
Radiotherapy related toxicity using CTC v5.0 (radiotherapy related acute and late toxicity) | Upto 2 years
  At baseline and at subsequent follow up till 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anil Tibdewal, Principal Investigator — Tata Memorial Hospital, Parel, Mumbai, Maharashtra, India
Locations (1):
- Tata Memorial Hospital, Parel, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No
Protocol manuscript is published and the results will be published in International peer-reviewed journal

REFERENCES:
- [Background] Tibdewal A, Agarwal JP, Srinivasan S, Mummudi N, Noronha V, Prabhash K, Patil V, Purandare N, Janu A, Kannan S. Standard maintenance therapy versus local consolidative radiation therapy and standard maintenance therapy in 1-5 sites of oligometastatic non-small cell lung cancer: a study protocol of phase III randomised controlled trial. BMJ Open. 2021 Mar 16;11(3):e043628. doi: 10.1136/bmjopen-2020-043628. PMID 33727268
- See also: Related Info — https://doi.org/10.1136/bmjopen-2020-043628